CLINICAL TRIAL: NCT01615575
Title: Transanal Haemorrhoidal Dearterialisation Versus Stapler Haemorrhoidopexy. A Randomized Trial With Long-term Follow-up
Brief Title: Transanal Haemorrhoidal Dearterialisation Versus Stapler Haemorrhoidopexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Erasmo Spaziani, PhD, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URomLS1
Record Dates: First submitted 2012-06-04; First posted 2012-06-08 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Haemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Haemorrhoidal dearterialisation (Active Comparator): Closure of the arterial blood flow to the haemorrhoidal plexus, using a dedicated proctoscope with a Doppler probe, and addiction of rectal mucopexy.
  Interventions: Procedure: Transanal haemorrhoidal dearterialisation
- Stapler haemorrhoidopexy (Active Comparator): Haemorrhoidopexy was performed with a single dedicated circular stapling device (PPH 03, Ethicon Endo-Surgery, Ohio, USA.)
  Interventions: Procedure: Stapler haemorrhoidopexy

INTERVENTIONS:
Procedure: Transanal haemorrhoidal dearterialisation — Closure of the arterial blood flow to the haemorrhoidal plexus, using a dedicated proctoscope with a Doppler probe, and a rectal mucopexy
  Arms: Haemorrhoidal dearterialisation
Procedure: Stapler haemorrhoidopexy — Haemorrhoidopexy with a single dedicated circular stapling device (PPH 03, Ethicon Endo-Surgery, Ohio, USA).
  Arms: Stapler haemorrhoidopexy

SUMMARY:
The aim of the present study was to compare the results of transanal haemorrhoidal dearterialisation and stapler haemorrhopidopexy in the treatment of grade III and IV haemorrhoids with a long-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* grade III and IV hemorrhoids requiring hemorrhoidectomy.

Exclusion Criteria:

* first and second degree hemorrhoids
* patients with firm and fibrotic external irreducible haemorrhoids
* thrombosed hemorrhoids; recurrent hemorrhoids after previous surgical treatment
* history of inflammatory bowel disease; history of colon, rectal or anal cancer
* inability to give informed consent
* age < 18 years
* pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Recurrence | 42 months
  A telephone interview with a structured questionnaire at a median follow-up of 42 months.

SECONDARY OUTCOMES:
Postoperative pain | 24 hr
  Pain score 24 hr after operation
Complications | One month
  Intra and postoperative complication within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Pierino Lucarelli, MD, FRCS, Principal Investigator
Locations (1):
- The City Hospital, Dubai, United Arab Emirates